CLINICAL TRIAL: NCT00624065
Title: COR111096, A Randomized, Double-Blind, Active-Controlled, Parallel Group, Multicenter Study Comparing the Proportion of Subjects With Stage 1 or 2 Essential Hypertension Who Achieve Target Blood Pressure While Receiving Either Carvedilol CR + Lisinopril or Lisinopril Monotherapy
Brief Title: Research Study To Test Carvedilol CR + Lisinopril Versus Lisinopril + Placebo In Patients With High Blood Pressure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COR111096
Record Dates: First submitted 2008-02-14; First posted 2008-02-26 (Estimated); Results first posted 2009-08-03 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-11

CONDITIONS: Hypertension
Keywords: target blood pressure; hypertension; COREG CR; carvedilol CR; Stage 1 or 2 essential hypertension; lisinopril
MeSH Terms: conditions — Hypertension | interventions — Lisinopril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- carvedilol CR + lisinopril (Experimental)
  Interventions: Drug: carvedilol controlled release/lisinopril
- lisinopril + placebo (Active Comparator)
  Interventions: Drug: lisinopril + placebo

INTERVENTIONS:
Drug: carvedilol controlled release/lisinopril — carvedilol CR + lisinopril given as separate pills
  Arms: carvedilol CR + lisinopril
Drug: lisinopril + placebo — lisinopril plus placebo to match carvedilol CR
  Arms: lisinopril + placebo

SUMMARY:
Randomized, double-blind, parallel group, multicenter study of subjects with Stage 1 or 2 essential hypertension who are not at target blood pressure (<140/90mmHg) at Baseline. Subjects will be randomized to receive either carvedilol CR + lisinopril or lisinopril + placebo. Subjects will be uptitrated over a 6 week period until target blood pressure (<140/90mmHg) is met. The primary objective of the study is to compare the proportion of subjects who achieve target blood pressure after 6 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18-80 years; stage 1 or 2 hypertension currently receiving 0 or 1 antihypertensive medication; mean sitting systolic blood pressure >/=140mmHg to </=170mmHg, or mean sitting diastolic blood pressure >/=90 to </=105mmHg. Subjects taking one hypertensive medication had their medication withdrawn and entered a wash-out phase prior to randomization.

Exclusion Criteria:

* Subject taking two or more antihypertensive medications, known contraindication to angiotensin-converting enzyme (ACE) inhibitors or alpha- or beta-blocker therapy, subject has Type 1 or Type 2 diabetes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (69):
- United States (69):
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Goodyear, Arizona
  - GSK Investigational Site, Litchifield Park/Arizona, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Beuna Park, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Poway, California
  - GSK Investigational Site, San Ramon, California
  - GSK Investigational Site, Tustin, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Tamarac, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, Aurora, Illinois
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Gillespie, Illinois
  - GSK Investigational Site, Elkhart, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Paducah, Kentucky
  - GSK Investigational Site, Slidell, Louisiana
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Butte, Montana
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, East Syracuse, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Westfield, New York
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Fargo, North Dakota
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Corvallis, Oregon
  - GSK Investigational Site, Altoona, Pennsylvania
  - GSK Investigational Site, Havertown, Pennsylvania
  - GSK Investigational Site, Jersey Shore, Pennsylvania
  - GSK Investigational Site, Lansdale, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Manning, South Carolina
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Georgetown, Texas
  - GSK Investigational Site, Grand Prairie, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Sugar Land, Texas
  - GSK Investigational Site, Draper, Utah
  - GSK Investigational Site, Magna, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Sandy City, Utah
  - GSK Investigational Site, Bellingham/Washington, Washington
  - GSK Investigational Site, Gig Harbor, Washington
  - GSK Investigational Site, Olympia, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Beloit, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] GSK has submitted manuscripts of these study results to peer-reviewed scientific journals which were not accepted for publication. GSK is providing the attached study results summary with a conclusion.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: COR111096 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: COR111096 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: COR111096 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: COR111096 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: COR111096 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: COR111096 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: COR111096 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Lisinopril: Lisinopril monotherapy (10, 20, or 40 mg once daily)
- Carvedilol CR + Lisinopril: Carvedilol controlled release (CR) + lisinopril (20 + 10, 20 + 20, or 40 + 20 mg once daily)
Period: Overall Study
Arm/Group | Lisinopril | Carvedilol CR + Lisinopril
Started | 216 | 216
Completed | 197 | 192
Not Completed | 19 | 24
Not completed — Adverse Event | 5 | 6
Not completed — Lost to Follow-up | 4 | 1
Not completed — Consent withdrawn | 6 | 5
Not completed — Lack of Efficacy | 0 | 3
Not completed — Met protocol-defined stopping criteria | 4 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lisinopril | Carvedilol CR + Lisinopril | Total
Number analyzed (Participants) | 216 | 216 | 432
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (11.9) | 54.1 (9.8) | 54.1 (10.9)
Gender [Count of Participants; unit: Participants]
  Female | 95 | 95 | 190
  Male | 121 | 121 | 242
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage (AA/AH) | 45 | 29 | 74
  American Indian or Alaska Native | 1 | 2 | 3
  Japanese/East Asian/South East Asian Heritage | 16 | 6 | 22
  Mixed Asian Heritage | 1 | 0 | 1
  White | 150 | 178 | 328
  AA/AH & American Indian or Alaska Native | 2 | 0 | 2
  AA/AH & American Indian or Alaska Native & White | 1 | 0 | 1
  AA/AH & White | 0 | 1 | 1
Baseline Blood Pressure [Mean (Standard Deviation); unit: mm/Hg]
  Baseline Sitting Systolic Blood Pressure (SBP) | 149.8 (10.25) | 148.8 (10.30) | 149.3 (10.27)
  Baseline Sitting Diastolic Blood Pressure (DBP) | 92.2 (8.12) | 92.2 (6.84) | 92.2 (7.50)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Mean Sitting Cuff Blood Pressure <140/90 mmHg at the End of 6 Weeks of Treatment
Description: Sitting cuff blood pressure was calculated as the mean of three measurements taken approximately 2 minutes apart, and before the morning dose.
Time Frame: Week 6
Population: Intent to Treat Efficacy (ITTE) Population: all randomized participants with efficacy (vital signs) data after a minimum of 4 weeks of treatment
Measure: Number; unit: Participants
Arm/Group | Lisinopril | Carvedilol CR + Lisinopril
Number analyzed (Participants) | 203 | 201
Participants
  Responders (mean BP <140/90 mmHg) | 139 | 137
  Non-responders (SBP >/=140 mmHg or DBP >/=90 mmHg) | 64 | 64
Statistical Analysis 1: Comparison: Lisinopril vs Carvedilol CR + Lisinopril; Test type: Superiority or Other; p = 0.8822, Regression, Logistic; Odds Ratio (OR) = 0.968, 95% CI [0.63 to 1.49]

2. Secondary Outcome: Mean Change From Baseline in Sitting Systolic Blood Pressure (sSBP) and Sitting Diastolic Blood Pressure (sDBP) at Week 6
Description: Mean change was calculated as Week 6 values minus Baseline values.
Time Frame: Baseline and Week 6
Population: ITTE
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lisinopril | Carvedilol CR + Lisinopril
Number analyzed (Participants) | 203 | 201
mmHg
  sSBP (mmHg) | -17.05 (12.27) | -16.07 (13.49)
  sDBP (mmHg) | -10.15 (7.52) | -9.14 (9.65)

ADVERSE EVENTS:
Description: The frequency threshold for reporting Other Adverse Events is 1% in either treatment group.
Arm/Group | Lisinopril | Carvedilol CR + Lisinopril
Serious Adverse Events (participants affected / at risk) | 2 | 3
Other Adverse Events (participants affected / at risk) | 50 | 54
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Lisinopril | Carvedilol CR + Lisinopril
Cardiac failure (Cardiac disorders) | 1/216 | 0/216
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0/216 | 1/216
Non-cardiac chest pain (General disorders) | 0/216 | 1/216
Meningitis viral (Infections and infestations) | 0/216 | 1/216
Overdose (Injury, poisoning and procedural complications) | 1/216 | 0/216
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/216 | 1/216
Headache (Nervous system disorders) | 0/216 | 1/216
Suicide attempt (Psychiatric disorders) | 1/216 | 0/216
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Lisinopril | Carvedilol CR + Lisinopril
Fatigue (General disorders) | 11/216 | 15/216
Cough (Respiratory, thoracic and mediastinal disorders) | 13/216 | 11/216
Headache (Nervous system disorders) | 11/216 | 10/216
Dizziness (Nervous system disorders) | 9/216 | 9/216
Nausea (Gastrointestinal disorders) | 6/216 | 5/216
Diarrhea (Gastrointestinal disorders) | 3/216 | 7/216
Arthralgia (Musculoskeletal and connective tissue disorders) | 4/216 | 2/216
Gastroenteritis (Infections and infestations) | 3/216 | 3/216
Upper respiratory tract infection (Infections and infestations) | 3/216 | 3/216
Flushing (Vascular disorders) | 3/216 | 2/216
Bronchitis (Infections and infestations) | 1/216 | 3/216
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 1/216 | 3/216
Oedema peripheral (General disorders) | 3/216 | 1/216
Sinusitis (Infections and infestations) | 0/216 | 4/216
Urinary tract infection (Infections and infestations) | 4/216 | 0/216
Dyspepsia (Gastrointestinal disorders) | 0/216 | 3/216
Rash (Skin and subcutaneous tissue disorders) | 3/216 | 0/216

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.